CLINICAL TRIAL: NCT05127733
Title: Online Cognitive Behavioural Therapy for Substance Use Disorder: The Impact of Peer Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Breaking Free Online (BFO) (Unknown); Community Addictions Peer Support Association (CAPSA) (Unknown)
Responsible Party: Principal Investigator, Lena Quilty, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 031/2020
Record Dates: First submitted 2021-10-14; First posted 2021-11-19 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Substance Use Disorders
Keywords: Cognitive behavioral therapy; Online treatment; Peer support
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online Cogntivie Behavioural Therapy (Experimental): Breaking Free Online (BFO) is an online intervention, supporting adults struggling with substance use. It provides psychoeducation and skills building exercises in CBT and compatible approaches. The intervention strategies contained within BFO are provided via a six-domain biopsychosocial model used in CBT. Each domain of the model corresponds to a module in the BFO program which contains psychoeducation and an 'action' strategy to facilitate behaviour change. Data captured at the baseline assessment is used by the program to provide feedback to the individual on their levels of functioning across the six domains. The program then guides the user to concentrate on intervention strategies for domains with the greatest level of impairment.
  All groups will receive 'clinical monitoring,' including biweekly study assessments during the acute treatment period and monthly assessments during the six month follow-up period.
  Interventions: Behavioral: Online Cognitive Behavioural Therapy
- Online Cognitive Behavioural Therapy Plus Individual Peer Support (Experimental): BFO delivered with peer support will comprise BFO with at least weekly contact with a peer with lived experience. Peer support workers will receive training on how to facilitate participant engagement with and progress through the BFO program, as well as a weekly session plan. As part of this training, peer support workers will be given their own access code to use BFO and be encouraged to use the program. Session One constitutes an initial orienting to the program. Subsequent sessions review each information and action strategy in the BFO program, with a series of prompts to guide peer support of this content.
  All groups will receive 'clinical monitoring,' including biweekly study assessments during the acute treatment period and monthly assessments during the six month follow-up period.
  Interventions: Behavioral: Online Cognitive Behavioural Therapy; Behavioral: Individual Peer Support
- Group Peer Support (Active Comparator): The control condition will consist of group peer support facilitated by trained peers and offered through the Community Addictions Peer Support Association (CAPSA). The group meets weekly and will offer participants a space to share their experiences and receive support.
  All groups will receive 'clinical monitoring,' including biweekly study assessments during the acute treatment period and monthly assessments during the six month follow-up period.
  Interventions: Behavioral: Group Peer Support

INTERVENTIONS:
Behavioral: Online Cognitive Behavioural Therapy — Interactive program utilizing cognitive behavioural therapy principles that guides users through its components and provides feedback, which facilitates behavior change (i.e., reduction in alcohol or substance use).
  Other Names: Breaking Free Online (BFO)
  Arms: Online Cognitive Behavioural Therapy Plus Individual Peer Support; Online Cogntivie Behavioural Therapy
Behavioral: Individual Peer Support — Weekly meetings with a trained peer support worker who guides participants through the BFO platform, reviews the platform's content with them, and supports them in the creation of an action strategy based on the platform's suggestions.
  Other Names: BFO Peer Support
  Arms: Online Cognitive Behavioural Therapy Plus Individual Peer Support
Behavioral: Group Peer Support — Meetings with a group of peers led by a trained peer support worker/volunteer which will offer the participants an opportunity to discuss their experiences in a supportive and open environment.
  Other Names: All People All Pathways
  Arms: Group Peer Support

SUMMARY:
The purpose of this study is to evaluate the efficacy and cost-effectiveness of Breaking Free Online, in a comparison of outpatients seeking treatment for substance use disorder who receive standard care with group peer support, versus with access to Breaking Free Online, versus with access to Breaking Free Online and individual peer support.

DETAILED DESCRIPTION:
A total of 225 outpatients receiving standard care for substance use disorder from the Centre for Addiction and Mental Health will be randomized to receive clinical monitoring (CM) with group peer support, Breaking Free Online only, or Breaking Free Online with individual peer support, in an eight-week trial with a six-month follow-up period. The primary outcome is substance use frequency; secondary outcomes include substance use problems, depression, anxiety, quality of life, treatment engagement, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and above
2. Fluency in English
3. Understanding and willingness to comply with study requirements & provide informed consent
4. Current substance use disorder
5. Have used alcohol or substances within the past 30 days
6. Registration with CAMH Addictions Program outpatient services

Exclusion Criteria:

1. Current psychosis or mania
2. Current psychiatric disorder requiring care more urgently than substance use, including acute intoxication or withdrawal requiring medical attention
3. Significant neurological disorder or physical illness likely to interfere with participants
4. Any known practical factors that would preclude participation (e.g., extended absences)
5. Inability to read at a sixth grade level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow-Back | 30 days
  Frequency (days) of substance use over the past 30 days

SECONDARY OUTCOMES:
Qualitative Interview | 10 months
  This interview will follow established principles of qualitative research and include questions specifically designed for this study. This interview will have a two-pronged focus including (1) barriers and facilitators to the implementation of online CBT and (2) a complementary ethnographic focus on "health work" patients engage in to understand the impact of online CBT and explore ways to optimally deliver support during the care journey. Thematic analysis of interview data will be undertaken to offer a summative description of how patients give meaning to their experience.
Program and Client Costs- Substance Abuse Treatment (PACC-SAT) | 7 days
  Healthcare costs
Severity of Dependence Scale | 1 month
  A self-report questionnaire assessing the severity of drug dependence. The minimum possible score is 0 and the maximum is 15, with higher scores indicating more severe dependence.
Alcohol Use Disorder Identification Test | 1 month
  Alcohol use and associated harms. The minimum possible score is 0 and the maximum is 40, with higher scores indicating more harmful alcohol use.
Drug Use Disorders Identification Test | 1 month
  Drug use and associated harms. The minimum possible score is 0 and the maximum is 44, with higher scores indicating more harmful drug use.
Patient Health Questionaire-9 | 14 Days
  Depression symptom severity. The minimum possible score is 0 and the maximum is 27, with higher scores indicating more severe depression.
Generalized Anxiety Disorder-7 | 14 days
  Generalized anxiety symptom severity. The minimum possible score is 0 and the maximum is 24, with higher scores indicating more severe anxiety.
World Health Organization Quality of Life Assessment | 4 weeks
  Quality of life over four domains. Subscale scores are calculated for 4 domains (physical health, psychological, social relationships and environment) and for "overall" and "general health" quality of life. Subscale scores have a range of 0 to 100, with higher scores indicating greater quality of life.
Substance Use Calendar (SUC) | 14 days
  This chart that will collect self-reports of alcohol and drug use and quantities of primary substance used.
Brief COPE Scale | Baseline, up to 8 weeks, and up to 6 months
  Frequency of use of different coping strategies in response to stressors. Each coping strategy is rated on a scale of 1 to 4, with higher scores indicating more use of the strategy.
Adult Hope Scale | Baseline, up to 8 weeks, and up to 6 months
  Assessment of level of hope. The minimum possible score is 12 and the maximum is 96, with higher scores indicating higher levels of hope.
Positive and Negative Affect Schedule - Expanded Form | 30 days
  Positive and negative affect as well as additional specific affects. The minimum score for each emotion is 1 and the highest possible score for each emotion is 5, with higher scores indicating more intensity of that emotion. Composite scores are computed for general positive and general negative affect, with a minimum total score of 10 and a maximum total score of 50 for each type, with higher scores indicating higher presence of that type of affect. Additional specific affect total scores are also computed with higher scores indicating more presence of the affect.
Contemplation Ladder | Baseline, up to 8 weeks, and up to 6 months
  Assessment of participant perspectives about changing substance use. The minimum score is 1 and the highest possible score is 10, with higher scores indicating more change in substance use.
Treatment Acceptability/Adherence Scale | Baseline, up to 8 weeks, and up to 6 months
  Treatment acceptability and anticipated or actual adherence in response to a given treatment. The minimum possible score is 10 and the maximum is 70, with higher scores indicating more acceptability or adherence to the treatment.
World Health Organization Disability Assessment Schedule 2.0 | 30 days
  Overall level of functioning. The minimum possible score is 0 and the maximum is 100, with higher scores indicating more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Lena C. Quilty, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Campbell Family Mental Health Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quilty LC, Wardell JD, Garner G, Elison-Davies S, Davies G, Klekovkina E, Corman M, Alfonsi J, Crawford A, de Oliveira C, Weekes J. Peer support and online cognitive behavioural therapy for substance use concerns: protocol for a randomised controlled trial. BMJ Open. 2022 Dec 12;12(12):e064360. doi: 10.1136/bmjopen-2022-064360. PMID 36523236
- See also: Description Information about research at the Centre for Addiction and Mental — http://www.camh.ca/research